CLINICAL TRIAL: NCT01939873
Title: A Prospective, Randomized, Controlled Trial
Brief Title: The Effect Of Kristeller Maneuver On Maternal And Neonatal Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kayseri Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Gökhan Açmaz, Kayseri Education and Research Hospital, Kayseri Education and Research Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Screening
Other Study IDs: KayseriERH
Record Dates: First submitted 2013-09-02; First posted 2013-09-11 (Estimated); Last update posted 2013-09-11 (Estimated); Status verified 2013-09

CONDITIONS: Secons Stage of Labor
Keywords: Kristeller maneuver; Second stage of labor;; Perineal laceration; Obstetrical outcome;; Neonatal outcome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- KRISTELLER (Experimental): Uterine fundal pressure
  Interventions: Behavioral: KRISTELLER
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: KRISTELLER
  Arms: KRISTELLER

SUMMARY:
The use of fundal pressure in management of the second stage of labor is controversial. The aim of this study is both to evaluate the effectiveness of fundal pressure in shortening the second stage of labor and to examine the related neonatal and maternal outcomes.

DETAILED DESCRIPTION:
Patients will be randomly allocated to two groups by using a computer-generated random number chart: Kristeller maneuver intervention (study) group (n=140) and control group (n=140). Umbilical artery blood gas will obtained to assess the newborn's acid-base status. The umbilical artery levels of creatinine kinase, creatinine kinase with myocardial specific isoform, aspartate amino transferase, alanine amino transferase, lactate dehydrogenase and lactic acid will be measured. Length of episiotomy and length of vagina will be measured at 45 degrees from the midline. Each patient's vaginal laceration, cervical laceration, length of episiotomy and vagina before and after delivery and duration of the second stage of labor in minutes will be recorded. Neonatal information will include: infant birth weight, apgar scores, babies requiring pediatric help, and admission of neonatal intensive care units.

ELIGIBILITY:
Inclusion Criteria:

* Pregnants who were administered for delivery and signed informed consent form were included into the study.

Exclusion Criteria:

* Pregnant who required oxytocin augmentation, multiple gestations, pregnant with medical problems (such as asthma, thyroid, cardiac, liver, kidney disease, preeclampsia and diabetes), pregnant with previous caesarean and pregnant whose estimated fetal weight <2500gr or >4000gr were not included into the study.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 285 (Actual)
Dates: Start 2012-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
vaginal laceration, cervical laceration, length of episiotomy and vagina before and after delivery | up to 6 months
  It is a composite outcome measure consisting of multiple measures.

SECONDARY OUTCOMES:
The umbilical artery levels of creatinine kinase, creatinine kinase with myocardial specific isoform, aspartate amino transferase, alanine amino transferase, lactate dehydrogenase and lactic acid were measured. | up to 6 months
  It is a composite outcome measure consisting of multiple measures.

CONTACTS AND LOCATIONS:
Locations (1):
- Gökhan, Kayseri, Turkey (Türkiye)